CLINICAL TRIAL: NCT02702310
Title: Prospective Observational Trial of Low-Dose Total Skin Electron Therapy in Mycosis Fungoides Using Rotisserie Technique
Brief Title: Low-Dose Total Skin Electron Therapy in Treating Patients With Refractory or Relapsed Stage IB-IIIA Mycosis Fungoides
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Austin Kirschner, Principal Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC RAD 1633; NCI-2015-02293 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Mycosis Fungoides; Refractory Mycosis Fungoides; Stage I Mycosis Fungoides; Stage II Mycosis Fungoides; Stage III Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Quality of Life/ Grading Skin Findings: Patients' baseline quality of life is established by completion of an initial questionnaire, and skin lesion burden is quantified by physical examination using a recommended system . Following the standard of care radiation therapy, patients' completion of questionnaire, and physical examination is repeated for continued assessment.
  Interventions: Other: Quality-of-Life Assessment; Other: Objective Grading of Skin Findings

INTERVENTIONS:
Other: Quality-of-Life Assessment — At initial visit (day 1) - for determination of a baseline quality of life, patients will be given a self-reported questionnaire called the Skindex-29. Following standard of care radiation treatments, at weeks 6 & 12, and every 3 months thereafter, patients will complete the Skindex-29 questionnaire.
Other: Objective Grading of Skin Findings — At initial visit (day 1) , using mSWAT the radiation oncologist can follow the patient's treatment response by accurately grading the severity of the patient's skin findings. Following standard of care radiation treatments, at weeks 6 & 12, and every 3 months thereafter, mSWAT will again be determined by physician. Follow-up visits will continue until patient has a change in disease.
  Other Names: Skindex-29 questionnaire

SUMMARY:
This clinical trial studies low- dose total skin electron therapy in treating patients with stage IB-IIIA mycosis fungoides that has not responded to previous treatment (refractory) or has returned after a period of improvement (relapsed). Radiation therapy uses high energy electrons to kill tumor cells and shrink tumors. Rotisserie technique is a method in which the patient receives total skin electron therapy while standing on a rotating platform. Giving low dose total skin electron therapy using rotisserie technique may kill tumor cells, while having fewer side effects, and may allow therapy to be repeated in future if clinically indicated.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the skin-related quality of life using an established method (Skindex-29), with comparisons made between pre-treatment and each of follow-up post-treatment skin assessments.

II. To assess the durability of response using an established method (modified Severity-Weight Assessment [mSWAT] tool), with comparisons made between pre-treatment and each of follow-up post-treatment skin assessments.

III. To determine side effect profile for low dose total skin electron therapy (TSE) for mycosis fungoides administered via rotisserie technique.

OUTLINE:

The investigational portion of this research study involves collecting quality of life (QOL) questionnaire data and objective measurements of patients' skin responses, which are obtained by the radiation oncologist during the patient's standard of care radiation treatment planning. Patients will also undergo standard of care low-dose total skin electron therapy for under 1 hour daily on days 10-21.

After completion of study treatment, patients are followed up at 6 and 12 weeks, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed mycosis fungoides stage IB-IIIA
* Skin manifestations of mycosis fungoides that are refractory to or have relapsed on at least one prior therapy, which may include topical steroids
* Life expectancy > 6 months

Exclusion Criteria:

* Serious medical condition that would make treatment unsafe
* Pregnant or lactating patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The high volume of cutaneous lymphoma patients seen at Vanderbilt makes it likely to significantly contribute to the knowledge about this treatment technique. Given the rarity of this disease, with Vanderbilt being a major treatment center for mycosis fungoides, the goal is to systematically contribute to the data for low-dose total skin electron therapy in order to prospectively assess these endpoints. It is expected to find skin manifestations of mycosis fungoides that are refractory or have relapsed on at least one prior therapy. Patients with prior skin electron therapy, including either high or low-dose total skin electron therapy, are permitted on this protocol if the radiation oncologist determines that low-dose radiation therapy can safely carried out. The goal is to assess quality of life and accurately grade skin findings following this non-experimental, standard of care, total skin electron radiation treatment.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-05-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in skin-related quality of life assessed by Skindex-29 | Baseline to up to 3 years
  Skindex-29 is a validated quality of life questionnaire to help quantify how mycosis fungoides may affect one's quality of life on a day to day basis, including emotional impact of the skin disease.

SECONDARY OUTCOMES:
Change in the durability of response assessed by mSWAT tool | Baseline to up to 3 years
  mSWAT is the Modified Severity Weighted Assessment Tool used by the radiation oncologist during complete physical examination to quantify skin findings of patches, plaques, and tumors in all regions of the body; this would help the radiation oncologist and dermatologist to better follow the response to treatment.
Incidence of side effects of low dose total skin electron therapy administered via rotisserie technique | Up to 3 years
  The patient will be closely monitored by the radiation oncologist during treatment, with at least 2-3 visits while patient is on treatment. Side effects will be documents in patient medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Kirschner, MD, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Newman NB, Patel CG, Ding GX, Zic JA, Zwerner J, Osmundson EC, Kirschner AN. Prospective observational trial of low-dose skin electron beam therapy in mycosis fungoides using a rotational technique. J Am Acad Dermatol. 2021 Jul;85(1):121-127. doi: 10.1016/j.jaad.2020.12.023. Epub 2020 Dec 14. PMID 33333150
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/